CLINICAL TRIAL: NCT02178631
Title: Effectiveness of Internet-based Depression Treatment (EVIDENT) in Severe Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Björn Meyer, Gaia AG, Hamburg, Germany / Department of Psychology, City University, London, United Kingdom (Unknown); University of Hamburg-Eppendorf (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Philipp Klein, Dr. med., University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVIDENTplus
Record Dates: First submitted 2014-06-25; First posted 2014-07-01 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Severe Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deprexis (Experimental): Online self-help
  Interventions: Behavioral: Deprexis
- CAU (Active Comparator): Care as usual
  Interventions: Other: CAU

INTERVENTIONS:
Behavioral: Deprexis — Online self-help
  Arms: Deprexis
Other: CAU — Care as usual
  Arms: CAU

SUMMARY:
Online self-help is an innovative way of providing self-help. The investigators want to study the effect of an interactive online self-help-program (Deprexis) in the treatment of severe depressive symptoms. Participants will be randomised to either twelve weeks of online-self help or a waiting-list control. Symptoms of depression and other aspects will be assessed over a six months period. The investigators hypothesise that online self-help is superior to the control condition in alleviating depressive symptoms and preventing full blown depression.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65, ability to read German, willingness to participate in a telephone diagnostic interview, achieving a score of at least 15 on the PHQ-9 in an initial screening, and providing written informed consent

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia or bipolar disorder (as determined by a telephone diagnostic interview) or current suicidality (as determined in a telephone interview)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 items (PHQ-9) | Change from Baseline to post (3mths).

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms - Self-Rreport (QIDS-SR16) | Baseline, post (3 mths), follow-up (6 mths)
Generalized Anxiety Disorder - 7 (GAD-7) | Baseline, post (3 mths), follow-up (6 mths)
Patient Health Questionnaire - 15 items (PHQ-15) | Baseline, post (3 mths), follow-up (6 mths)
Short Form Health Survey - 12 (SF-12) | Baseline, post (3 mths), follow-up (6 mths)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (3):
  - Department of Psychiatry and Psychotherapy, University of Hamburg, Hamburg
  - Gaia AG, Hamburg
  - Department of Psychiatry and Psychotherapy, University of Luebeck, Lübeck
- Department of Clinical Psychology and Psychotherapy, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Klein JP, Berger T, Schroder J, Spath C, Meyer B, Caspar F, Lutz W, Greiner W, Hautzinger M, Rose M, Grafe V, Hohagen F, Andersson G, Vettorazzi E, Moritz S. The EVIDENT-trial: protocol and rationale of a multicenter randomized controlled trial testing the effectiveness of an online-based psychological intervention. BMC Psychiatry. 2013 Sep 28;13:239. doi: 10.1186/1471-244X-13-239. PMID 24074299
- [Derived] Kaiser T, Boschloo L, Berger T, Meyer B, Spath-Nellissen C, Schroder J, Hohagen F, Moritz S, Klein JP. Maintaining Outcomes of Internet-Delivered Cognitive-Behavioral Therapy for Depression: A Network Analysis of Follow-Up Effects. Front Psychiatry. 2021 Apr 20;12:598317. doi: 10.3389/fpsyt.2021.598317. eCollection 2021. PMID 33959044